CLINICAL TRIAL: NCT05667623
Title: A Multinational, Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Comparison Trial to Demonstrate the Superiority of 1% OPA-15406 Ointment to the Vehicle in Adult Patients With Atopic Dermatitis
Brief Title: To Demonstrate the Superiority of IMP (1% OPA-15406 Ointment) to the Vehicle in Adult Patients With AD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271-403-00014
Record Dates: First submitted 2022-12-02; First posted 2022-12-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1% OPA-15406 Ointment (Experimental): The 1% formulation of OPA-15406 ointment will be administered twice-daily (approximately 12 hours apart between morning and night administration) for 4 weeks/24 weeks. The amount of IMP (g) per dose is 10 g/m2 BSA and calculated.
  Interventions: Drug: 1% OPA-15406 Ointment
- 0% OPA-15406 Vehicle (Placebo Comparator): The vehicle of OPA-15406 vehicle will be administered twice-daily (approximately 12 hours apart between morning and night administration) for 4 weeks/24 weeks. The amount of IMP (g) per dose is 10 g/m2 BSA and calculated.
  Interventions: Other: 0% OPA-15406 Vehicle

INTERVENTIONS:
Drug: 1% OPA-15406 Ointment — Twice-daily administration for 4 weeks/24 weeks.
  Other Names: 0% OPA-15406 Vehicle
  Arms: 1% OPA-15406 Ointment
Other: 0% OPA-15406 Vehicle — Twice-daily administration for 4 weeks/24 weeks.
  Arms: 0% OPA-15406 Vehicle

SUMMARY:
This is a multinational (China and Korea), multicenter, randomized, double-blind, vehicle-controlled, parallel-group, comparison trial to demonstrate the superiority of 1% OPA-15406 ointment to the vehicle in adult AD subjects.

DETAILED DESCRIPTION:
1. Screening period After obtaining informed consent, the investigator will perform a screening examination. The screening period is defined as the period between the day of obtaining informed consent and the day of baseline visit (0 - 30 days).
2. Assessment period (4 weeks double blind treatment period) The assessment period is defined as the period between the day of baseline visit and the end of Week 4 visit (or the end of withdrawal visit). The subject who meets the inclusion criteria and does not meet the exclusion criteria at the baseline visit will be allocated to the 1% formulation of OPA-15406 or the comparator (vehicle [placebo]). The allocated IMP will be administered to the treatment area from the day of baseline visit twice-daily for 4 weeks. After the baseline visit, the examinations will be performed at Weeks 1, 2, and 4. If a subject discontinues the IMP administration between the day of baseline visit and the day of Week 4 visit, a withdrawal visit will be performed for that subject.
3. 4 Weeks Double Blind The trial period for individual subject is the period from the day of obtaining the subject's written informed consent to the day of the Week 4 visit or withdrawal visit. For subjects who missed the Week 4 visit or withdrawal visit, the day of discontinuation will be the day when the investigator determined that the subject was to be withdrawn from the trial. It does not include the follow-up period for AE.To evaluate the efficacy (secondary endpoint) and safety of IMP (1% OPA-15406 ointment) when administered twice-daily for 4 weeks in adult patients with AD.
4. 24 Weeks Open label, long term treatment period (China only) To be eligible for long term treatment, subjects must complete the randomized, double-blind treatment. Subjects must be judged by their investigators to have the potential for clinical benefit by longer-term exposure to OPA-15406, they can continue to receive 1% OPA-15406 open treatment for up to 24 weeks based on the informed consent of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization status: Outpatient.
2. Age: 15 to 70 years old, inclusive (at time of obtaining informed consent), either male or female (only for 4 weeks double blind treatment).
3. Able to provide written informed consent. For subjects under 18 years old (Korea: 19 years old), written informed consent must be obtained from both the subject and the subject's legal guardian.
4. Diagnosis of AD based on the criteria of Hanifin and Rajka. (See Appendix 1).
5. History of AD for at least 3 years.
6. Atopic dermatitis affecting ≥5% to ≤40% of BSA (excluding scalp) at the screening and baseline visit (only for 4 weeks double blind treatment).
7. IGA score of 2 or 3 at the screening and baseline visit (only for 4 weeks double blind treatment).

Exclusion Criteria:

1. Subjects who are pregnant, possibly pregnant, or breastfeeding, who desire to become pregnant or to have their partner become pregnant during the trial period and up until 30 days after the final administration of IMP, or who are unable to either remain abstinent or employ at least two of the specified birth control methods (vasectomy, tubal ligation, vaginal diaphragm, intrauterine device [IUD], birth control pill, condom with spermicide, etc.) during the trial period and up until 30 days after the final administration of IMP.
2. Subjects who defined as AD or contact dermatitis rapid deterioration, within 28 days prior to the baseline visit.
3. Subjects who have a concurrent or history of skin disease other than AD (e.g., acne, psoriasis, etc.) and who are judged inappropriate for assessment of AD in the present trial.
4. Subjects who have an active viral skin infection (e.g., herpes simplex, herpes zoster, chicken pox) or clinical signs of such infection.
5. Subjects with a current or history of malignancy within the previous 5 years.
6. Subjects with a current or history of recurrent bacterial infection resulting in hospitalization or requiring intravenous antibiotic treatment within the past 2 years.
7. Subjects with a clinically significant complication or history of any of the following disorders that the investigator judges would prevent safe conduct of the trial or impact efficacy assessment of the IMP:

   * Cardiac disease (e.g., rheumatic fever or heart valve replacement).
   * Endocrinologic disease (e.g., severe or uncontrolled diabetes).
   * Pulmonary disease.
   * Neurologic disease.
   * Psychiatric disease.
   * Hepatic disease (e.g., carriers of hepatitis B, hepatitis C, etc.).
   * Renal disease.
   * Hematologic disease.
   * Immunologic or immunocompromised disease (e.g., acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome, carriers of human immunodeficiency virus [HIV] antibodies, etc.).
   * Other major disease (e.g., systemic fungal infection) or other severe uncontrolled condition (e.g., drug or alcohol abuse) judged by the investigator to pose a health risk to the subject or to have the potential to impact efficacy assessment of the IMP.
8. Subjects with any of the following hematology or serum chemistry results at screening visit:

   * White blood cell count: ≤3, 000/µL (3 ×109/L) or >14, 000/µL (14 ×109/L).
   * Platelets: ≤100, 000/µL (100 ×109/L).
   * Hemoglobin: <9 g/dL (90 g/L).
   * Serum creatinine: ≥2 mg/dL (176.8 μmol/L).
   * Aspartate aminotransferase (AST) (glutamic oxaloacetic transaminase [GOT]): >2 × ULN.
   * Alanine aminotransferase (ALT) (glutamic pyruvic transaminase [GPT]): >2× ULN.
   * Total bilirubin: ≥2.0 mg/dL (34.2 μmol/L).
   * Any other abnormal laboratory test result that the investigator judges to be a clinically significant abnormality.
9. Subjects who are judged by the investigator to have a clinically significant abnormal blood pressure or pulse rate at the screening and baseline visits.
10. Subjects who are unable to stop allergen immunotherapy (or desensitization therapy) from 3 months prior to providing informed consent until the Week 4 visit (or at the time of withdrawal visit).
11. Subjects who are unable to stop treatment with ultraviolet A, narrowband ultraviolet B, and ultraviolet B from 28 days prior to the baseline examination until the Week 4 visit/ 24 weeks (long-term administration).
12. Subjects who are unable to stop using systemic corticosteroids, systemic immunosuppressant's, systemic antimetabolites, systemic retinoid, and biologics from 28 days prior to the baseline visit until the Week 4 visit/ 24 weeks (long-term administration).
13. Subjects who are unable to stop using topical corticosteroids for skin (excluding scalp) categorized as very strong potency in Appendix 2 'Rank of Topical Corticosteroids' from 21 days prior to the baseline visit until the Week 4 visit/ 24 weeks (long-term administration).
14. Subjects who are unable to stop using topical corticosteroids for skin (excluding scalp) categorized as strong potency in Appendix 2 'Rank of Topical Corticosteroids', topical corticosteroids other than those for skin, topical immunosuppressant's, topical retinoid, topical antihistamine and topical non-steroidal anti-inflammatory drugs (excluding for scalp) from 7 days prior to the baseline visit until the Week 4 visit/ 24 weeks (long-term administration). However, intra-ocular, intra-nasal, intra-auricular, and inhaled corticosteroids may be considered if the investigator judges that their use will not impact assessment of the affected area.
15. Subjects who are unable to stop using topical corticosteroids for skin (excluding scalp) categorized as low or medium potency in Appendix 2 'Rank of Topical Corticosteroids' from 4 days prior to the baseline visit until the Week 4 visit/ 24 weeks (long-term administration).
16. Subjects who are unable to continue in the trial without changing the dosage and administration of systemic antihistamines, sodium cromogicate, tranilast, or suplatast tosilate from 7 days prior to the baseline visit until the Week 4 visit/ 24 weeks (long-term administration).
17. Subjects with known hypersensitivity (including history) to any drugs (prescription, OTC, etc.) or any ingredient of OPA-15406 ointment (e.g., white petrolatum, mineral oil, paraffin, white wax, or propylene carbonate).
18. Subjects with known plans to receive any of the prohibited concomitant drugs or therapies during the trial period.
19. Subjects who have participated in previous trials for OPA-15406 and have been administered the IMP (only for 4 weeks double blind treatment).
20. Subjects who have used any other investigational drug within 4 months prior to the baseline visit or who are scheduled to participate in any other clinical trial during the trial period.
21. Subjects who have never been treated with medication for AD or who are satisfied with their current AD treatment regimen.
22. Subjects who do not respond at all to treatment with existing topical drugs for AD.
23. Subjects who are judged by the investigator to be inappropriate to participate in the trial for any other reason.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Success rate in Investigator's Global Assessment at Week 4 | 4 weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the percentage of subjects with Investigator's Global Assessment score of 0 or 1 with improvement by at least 2 grades. Subjects with missing Investigator's Global Assessment data will be handled as non-responders.

SECONDARY OUTCOMES:
Change from baseline in Investigator's Global Assessment at Week 4 | 4 weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the change from baseline in Investigator's Global Assessment at Week 4.
Success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index) and at Week 4 | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index) at Week 4.
Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index) at week 4 | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index) and at Week 4.
Eczema Area and Severity Index 50 (improvement of ≥50% in Eczema Area and Severity Index) at week 4 | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 50 (improvement of ≥50% in Eczema Area and Severity Index) and at Week 4.
Change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score at Week 4 | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score at Week 4.
Change from baseline in Verbal Rating Scale for Pruritus at Week 4 | 4 weeks
  The Verbal Rating Scale measures the intense pruritus in the past 24 hours following Verbal Rating Scale criteria( 0: None,1: Mild, 2: Moderate, 3: Severe). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by Change from baseline in Verbal Rating Scale (VRS) for Pruritus at Week 4
Change from baseline in Verbal Rating Scale for pruritus up to Day 7 | 7 Days
  The Verbal Rating Scale measures the intense pruritus in the past 24 hours following Verbal Rating Scale criteria( 0: None,1: Mild, 2: Moderate, 3: Severe). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's/subjects' judgment.
  The efficacy is assessed by Change from baseline in Verbal Rating Scale for Pruritus up to day 7.
Change from baseline in the total score of Patient-Oriented Eczema Measure at Week 4 | 4 weeks
  Eczema will be evaluated according to Patient-Oriented Eczema Measure .The subjects will answer 7 questions and describe their eczema. The investigator will confirm their responses and record the results in the source document and CRF. The total score of POEM is 28 points at the most. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by Change from baseline in the total score of Patient-Oriented Eczema Measure at Week 4
Change from baseline in the total score of Dermatology Life Quality Index at week 4 | 4 weeks
  The effects of symptoms on daily life will be evaluated according to Dermatology Life Quality Index (.The subjects will answer a total of 10 questions and describe the effects of the symptoms on their daily life (scale: symptoms, emotions, and functioning). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by change from baseline in the total score of Dermatology Life Quality Index at week 4.
Change from baseline in the total affected Body Surface Area (percent) at Week 4 | 4 weeks
  The efficacy is assessed by change from baseline in the total affected Body Surface Area (percent) at Week 4.
Success rate in Investigator's Global Assessment at Week 24 | 24 weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the percentage of subjects with Investigator's Global Assessment score of 0 or 1 with improvement by at least 2 grades. Subjects with missing Investigator's Global Assessment data will be handled as non-responders.
Time to IGA response | 24 weeks
  How long the subject's Investigator's Global Assessment score (IGA score of 0 or 1) improvement by at least 2 grades will take;
Success rate in EASI 75 (improvement of≥ 75% in EASI), EASI 90 (improvement of≥ 90% in EASI) and EASI 50 (improvement of≥ 50% in EASI) | 24 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index) , Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index), Eczema Area and Severity Index 500 (improvement of ≥50% in Eczema Area and Severity Index) at Week 24.
Changes from baseline in IGA score | 24 weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the change from baseline in Investigator's Global Assessment at Week 24.
Changes from baseline in the total score of EASI and each clinical sign score | 24 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score at Week 24.
Changes from baseline in the total score of Patient-Orientaed Eczema Measure (POEM) | 24 weeks
  Eczema will be evaluated according to Patient-Oriented Eczema Measure .The subjects will answer 7 questions and describe their eczema. The investigator will confirm their responses and record the results in the source document and CRF. The total score of POEM is 28 points at the most. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by Change from baseline in the total score of Patient-Oriented Eczema Measure at Week 24
Changes from baseline in the total affected BSA (%) | 24 weeks
  The efficacy is assessed by change from baseline in the total affected Body Surface Area (percent) at Week 24.

OTHER OUTCOMES:
Adverse events | 4 weeks/24 weeks
  Adverse events will be examined by frequency, severity, seriousness, discontinuation, and relationship to treatment.
Plasma concentrations of OPA-15406 | Week 4
  prior to IMP administration and 2 hours, 4 hours, and 8 hours postdose at Week 4(only in China)
Clinical laboratory tests | 4 weeks/24 weeks
  For each parameter (Hematology, Serum chemistry, Urine and/or serum pregnancy for women of childbearing potential), the descriptive statistics will becalculated for measured values and changes from the baseline at each visit for all subjects by treatment group. For qualitative urinalysis values of clinical laboratory tests, a shift table at each visit against the baseline will be created for all subjects.
Vital Signs | 4 weeks/24 weeks
  The number and percentage of subjects with potential clinical significant changes in body temperature, blood pressure (systolic and diastolic), and pulse rate will be calculated for all subjects.
Body Weigh | 4 weeks/24 weeks
  For each parameter and body weight, the descriptive statistics will be calculated for measured values and changes from baseline at each visit for all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, PHD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No